CLINICAL TRIAL: NCT04939415
Title: Multicenter Double Blind, Placebo Controlled RCT of Modified Qing Fei Pai Du Tang (mQFPD) for COVID-19
Brief Title: RCT of Modified Qing Fei Pai Du Tang (mQFPD) for COVID-19
Acronym: MACH19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Gordon Saxe, Director, Krupp Center for Integrative Research, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200633-1b
Record Dates: First submitted 2021-06-21; First posted 2021-06-25 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- modified Qing Fei Pei Du Tang (Experimental): encapsulated modified Qing Fei Pai Du Tang
  Interventions: Drug: mQFPD
- Placebo (Placebo Comparator): Organic brown rice
  Interventions: Drug: organic brown rice

INTERVENTIONS:
Drug: mQFPD — The dosage of mQFPD is 8 capsules three times a day for 14 consecutive days. It does not need to be consumed with food. It is best taken at least 30 minutes before OR at least 60 minutes after meals, in the morning, noon and evening. Accidentally missed doses will not need to be taken at a later time but will be recorded in a daily diary.
  Arms: modified Qing Fei Pei Du Tang
Drug: organic brown rice — The dosage of mQFPD is 8 capsules three times a day for 14 consecutive days. It does not need to be consumed with food. It is best taken at least 30 minutes before OR at least 60 minutes after meals, in the morning, noon and evening. Accidentally missed doses will not need to be taken at a later time but will be recorded in a daily diary.
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled clinical trial to evaluate a 21-herb formula named modified Qing Fei Pai Du Tang (mQFPD) to treat COVID-19-positive outpatients with mild-to-moderate symptoms assigned to self-quarantined and home management. This the study aims to establish the safety and feasibility of the use of mQFPD vs placebo in 66 total subjects. Subsequent trials will evaluate other therapeutics as well as the efficacy of mQFPD in a larger study population.

DETAILED DESCRIPTION:
Study participants will be assigned to one of two groups, either placebo or mQFPD. Participants will be screened and consented remotely. Both groups will receive blood draws at days 1 and 14, and will be sent study medication directly to their home from the investigational pharmacy. Baseline and end-of-study laboratory draws will be done at home via mobile phlebotomy. Adverse events and symptoms scores will be monitored by entry into a daily diary along with regular phone calls with the study coordinators.

At the end of the study, safety will be assessed by laboratory measures and adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

* Positive COVID-19 diagnosis within the prior 72 hours or within 9 days of symptom onset
* Age 18 years and older
* Women of childbearing potential must have a negative urine or serum hCG.
* Women of childbearing potential must have a negative serum pregnancy test at screening and agree to use contraception throughout the study period.
* Capable of documenting vitals, symptoms, and study product intake daily and communicating this information to the study team
* Willing to try to minimize alcohol, cannabis, and dairy products during the study period.

Exclusion Criteria:

1. Any of the following symptoms which, according to the CDC, require hospitalization:

   1. Trouble breathing
   2. Persistent pain or pressure in the chest
   3. New confusion or inability to arouse
   4. Bluish lips or face
2. Current use of investigational agents to prevent or treat COVID-19
3. Known liver disease (ALT/AST >3x ULN or diagnosis of cirrhosis)
4. Known renal disease (eGFR < 60 ml/min) or acute nephritis.
5. Uncontrolled hypertension (SBP>140 or DBP>90 while on medications)
6. Allergy to tree nuts
7. Bleeding dyscrasia or on anticoagulation (aspirin and/or clopidogrel is allowed)
8. Pregnant or breastfeeding women
9. Use of Tolbutamide
10. Use of systemic corticosteroids (hydrocortisone, cortisone, prednisolone, betamethasone, methylprednisolone, prednisone, dexamethasone). Inhaled budesonide is to be allowed.
11. Use of digoxin
12. Use of Oxacillin
13. Use of Interferon
14. Use of Vincristine
15. Use of Cyclosporine
16. Use of Amiodarone
17. Patients with a past medical history of epilepsy
18. Use of monoamine oxidase inhibitors (MAOI)
19. Use of Methamphetamine within the prior 30 days
20. Use of Cocaine within the prior 30 days
21. Use of aminoglycosides, carbamazepine, flecainide, lithium, phenytoin, phenobarbital, rifampicin, theophylline and warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Saxe, MD, Study Chair — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Started | 25 | 28
Completed | 24 | 23
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (13.5) | 43.0 (14.0) | 44.13 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 18 | 21 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 23 | 47
Total Protein Normal [Count of Participants; unit: Participants] | 22 | 22 | 44
Albumin Normal [Count of Participants; unit: Participants] | 22 | 22 | 44
Alkaline Phosphatase Normal [Count of Participants; unit: Participants] | 23 | 21 | 44
AST Normal [Count of Participants; unit: Participants] — aspartate aminotransferase
  Participants | 21 | 22 | 43
ALT Normal [Count of Participants; unit: Participants] — alanine transaminase
  Participants | 21 | 21 | 42
Total Bilirubin Normal [Count of Participants; unit: Participants] | 24 | 23 | 47
eGFR Normal [Count of Participants; unit: Participants] — estimated glomerular filtration rate
  Participants | 20 | 20 | 40
Prothrombin Time Normal [Count of Participants; unit: Participants] | 14 | 18 | 32
APTT Normal [Count of Participants; unit: Participants] — Activated partial thromboplastin time Population: APTT values were not available for all subjects.
  Participants
    number analyzed (Participants) | 23 | 22 | 45
    (all) | 21 | 16 | 37
ESR Normal [Count of Participants; unit: Participants] — Erythrocyte sedimentation rate
  Participants | 11 | 12 | 23
CRP Normal [Count of Participants; unit: Participants] — C-Reactive Protein Population: CRP values were not available for all participants.
  Participants
    number analyzed (Participants) | 22 | 23 | 45
    (all) | 14 | 12 | 26
LDH Normal [Count of Participants; unit: Participants] — Lactate dehydrogenase
  Participants | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Total Protein Normal to Abnormal Transition
Description: The Normal to Abnormal percentage reflects the percentage of participants with normal values at Day 1 that became abnormal at Day 14 relative to all participants with normal values at baseline.
Time Frame: 14 days
Population: Number of participants who were normal at baseline. Participants who were abnormal at baseline were excluded, therefore the number of participants in this analysis is different from the total number of participants in the mQFPD or Placebo groups described in the study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 22 | 22
percentage of participants | 4.5 | 4.6
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 1.000, Chi-squared, Corrected; ratio of frequencies = 0.000 — The Chi-square metric represents the difference between the expected and observed frequencies of an event, therefore it is the ratio of frequencies

2. Primary Outcome: Albumin Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 22 | 22
percentage of participants | 4.5 | 0.0
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 1.000, Chi-squared, Corrected; ratio of frequencies = 1.023 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Alkaline Phosphatase Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: Chi-square statistic could not be computed because all participants who were normal at baseline were also normal at day 14.
  Number of participants who were normal at baseline. Participants who were abnormal at baseline were excluded, therefore the number of participants in this analysis is different from the total number of participants in the mQFPD or Placebo groups described in the study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 23 | 21
percentage of participants | 0 | 0

4. Primary Outcome: AST Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 21 | 22
percentage of participants | 4.8 | 0
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.488, Chi-squared, Corrected; ratio of frequencies = 1.073 — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: ALT Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 21 | 21
percentage of participants | 9.5 | 0
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.488, Chi-squared, Corrected; ratio of frequencies = 2.10 — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Bilirubin Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
percentage of participants | 0 | 0

7. Primary Outcome: Adj. EGFR Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 20 | 20
percentage of participants | 15.0 | 0
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.231, Chi-squared, Corrected; ratio of frequencies = 3.243 — [estimate comment as in outcome 1, analysis 1]

8. Primary Outcome: Prothrombin Time Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 14 | 18
percentage of participants | 7.1 | 5.6
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 1.000, Chi-squared, Corrected; The Chi-square metric represents the difference between the expected and observed frequencies of an event, therefore it is the ratio of frequencies; ratio of frequencies = 0.034

9. Primary Outcome: APTT Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 21 | 16
percentage of participants | 9.5 | 12.5
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Other; p = 1.000, Chi-squared, Corrected; [statistical method as in outcome 8, analysis 1]; ratio of frequencies = 0.083

10. Primary Outcome: ESR Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 11 | 12
percentage of participants | 0 | 0

11. Primary Outcome: CRP Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: Number of participants who were normal at baseline. Participants who were abnormal at baseline were excluded.
  Number of participants who were normal at baseline. Participants who were abnormal at baseline were excluded, therefore the number of participants in this analysis is different from the total number of participants in the mQFPD or Placebo groups described in the study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 14 | 12
percentage of participants | 0 | 8.3
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.462, Chi-squared, Corrected; ratio of frequencies = 1.213 — [estimate comment as in outcome 1, analysis 1]

12. Primary Outcome: LDH Normal to Abnormal Transition
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 10 | 12
percentage of participants | 50 | 41.7
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 1.000, Chi-squared, Corrected; ratio of frequencies = 0.153 — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Mid-turbinate SARS CoV-2 Viral Load
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by changes in the SARS CoV-2 viral loads among mid-turbinate nasal swabs taken on days 0, 7 and 14.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: copies per mL
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
copies per mL
  Baseline (Day 1) | 17.9358 (7.07254) | 15.5282 (6.19859)
  Day 7 | 33.9909 (8.67777) | 32.7374 (8.62281)
  Day 14 | 37.5100 (5.05021) | 35.8814 (6.33340)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.668, Mixed Models Analysis; Group by Day interaction; F value = 0.185

14. Secondary Outcome: Albumin
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the Albumin of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
U/L
  Baseline (Day 1) | 4.43 (0.38) | 4.5 (0.22)
  Day 14 | 4.49 (0.37) | 4.56 (0.24)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.860, Mixed Models Analysis; F value = 0.032 — Group by Day interaction

15. Secondary Outcome: Alkaline Phosphatase
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the Alkaline Phosphatase of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
U/L
  Baseline (Day 1) | 83.96 (52.27) | 78.83 (24.03)
  Day 14 | 79.71 (26.31) | 75.32 (21.12)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.853, Mixed Models Analysis; F value = .035 — Group by Day interaction

16. Secondary Outcome: AST
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the AST of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
U/L
  Baseline (Day 1) | 28.54 (16.72) | 21.00 (7.32)
  Day 14 | 25.88 (10.84) | 17.91 (4.51)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.995, Mixed Models Analysis; F value = 0.000 — group by day interaction

17. Secondary Outcome: ALT
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the ALT of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
U/L
  Baseline (Day 1) | 28.46 (16.64) | 23.78 (17.18)
  Day 14 | 29.46 (17.73) | 19.41 (8.38)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.266, Mixed Models Analysis; F value = 1.27

18. Secondary Outcome: Total Bilirubin
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the Total Bilirubin of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
mg/dL
  Baseline (Day 1) | 0.39 (0.20) | 0.41 (0.20)
  Day 14 | 0.52 (0.20) | 0.42 (0.14)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.039, Mixed Models Analysis; F value = 4.533 — group by day interaction is reported
Statistical Analysis 2: Comparison: Modified Qing Fei Pei Du Tang; day 0 to day 14 for the mQFPD group were examined; Test type: Superiority; p < 0.001, ANOVA; Degrees of freedom: 1,23; F Ratio = 13.897
Statistical Analysis 3: Comparison: Placebo; day 0 to day 14 for the Placebo Group were examined; Test type: Superiority; p = 0.529, ANOVA; degrees of freedom: 1,20; F ratio = 0.410

19. Secondary Outcome: Adj. EGFR
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the Adj. EGFR of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
mL/min
  Baseline (Day 1) | 111.25 (24.90) | 117.09 (26.97)
  Day 14 | 107.65 (22.82) | 114.16 (27.72)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.710, Mixed Models Analysis; ratio of frequencies = .140 — group by day interaction

20. Secondary Outcome: Prothrombin Time
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the Prothrombin Time of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
sec
  Baseline (Day 1) | 11.88 (1.12) | 11.66 (1.15)
  Day 14 | 11.9 (1.02) | 11.28 (1.13)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.099, Mixed Models Analysis; F value = 2.855 — group by day interaction

21. Secondary Outcome: APTT
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the APTT of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
sec
  Baseline (Day 1) | 32.85 (6.01) | 33.37 (2.93)
  Day 14 | 32.24 (5.34) | 32.36 (2.94)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.228, Mixed Models Analysis; F value = 1.497 — group by day interaction

22. Secondary Outcome: INR
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the INR (international normalized ratio) of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients). The INR is a result of a blood test that measures how long it takes for blood to clot, also known as the prothrombin time (PT). The INR is calculated by comparing the PT to the mean normal prothrombin time (MNPT). Higher INR is thought to indicate liver dysfunction.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
ratio
  Baseline (Day 1) | 1.06 (0.10) | 1.1 (0.11)
  Day 14 | 1.07 (0.08) | 1.07 (0.11)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.119, Mixed Models Analysis; F value = 2.537 — group by day interaction

23. Secondary Outcome: ESR
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the ESR of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
mm/hr
  Baseline (Day 1) | 16.18 (11.56) | 18.80 (12.89)
  Day 14 | 12.50 (9.07) | 15.62 (17.19)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.643, Mixed Models Analysis; F value = .219 — group by day interaction

24. Secondary Outcome: CRP
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the CRP of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
mg/dL
  Baseline (Day 1) | 1.87 (5.01) | 0.88 (1.02)
  Day 14 | 1.10 (2.85) | 0.35 (0.25)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.817, Mixed Models Analysis; F value = .054

25. Secondary Outcome: LDH
Description: A secondary exploratory objective will be to evaluate COVID-19 severity among subjects in each of the two medication arms, compared with placebo, as ascertained by comparing the LDH of baseline laboratory data with end-of-treatment labs or on hospital admission labs (for hospitalized patients).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
U/L
  Baseline (Day 1) | 208.5 (80.95) | 177.48 (27.8)
  Day 14 | 210.29 (58.62) | 186.59 (24.68)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = 0.578, Mixed Models Analysis; F value = .315 — group by day interaction

26. Secondary Outcome: Symptom Count
Description: Symptom severity was assessed via a daily questionnaire across Days 0-14, where participants rated their symptoms on a scale of 0 (none or absent) to 3 (severe). A composite measure was created for each day, based on the 12 symptoms most commonly associated with COVID-19 (fever, fatigue, muscle aches, shortness of breath, shortness of breath upon exertion, cough, sore throat, stuffy nose, runny nose, loss of taste, loss of smell, headache), and counting the total number of symptoms present.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: Total Number of Symptoms
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
Total Number of Symptoms
  Baseline (Day 0) | 8.3750 (2.01759) | 7.3043 (2.49426)
  Day 1 | 7.5000 (2.82843) | 5.7826 (3.19028)
  Day 2 | 6.6667 (2.35292) | 6.0435 (2.24577)
  Day 3 | 6.3750 (2.65088) | 5.6522 (2.32787)
  Day 4 | 5.6667 (2.89928) | 5.1739 (2.53435)
  Day 5 | 5.3333 (2.85393) | 4.3043 (2.94549)
  Day 6 | 4.5000 (2.70266) | 3.9565 (2.93069)
  Day 7 | 4.5000 (2.53669) | 3.3043 (3.05160)
  Day 8 | 4.0833 (2.73332) | 2.9565 (2.63677)
  Day 9 | 3.9583 (2.85107) | 2.6522 (2.44222)
  Day 10 | 3.6667 (2.72934) | 2.3043 (2.26505)
  Day 11 | 3.2083 (2.35869) | 1.9545 (2.05814)
  Day 12 | 2.5417 (2.50181) | 1.6364 (2.03646)
  Day 13 | 2.6250 (2.46387) | 1.6818 (1.83579)
  Day 14 | 2.3750 (2.49891) | 1.8182 (1.96726)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = .643, Mixed Models Analysis; F value = .215 — day by group interaction

27. Secondary Outcome: Symptom Severities
Description: Symptom severity was assessed via a daily questionnaire across Days 0-14, where participants rated their symptoms on a scale of 0 (none or absent) to 3 (severe). A composite measure was created for each day, based on the 12 symptoms most commonly associated with COVID-19 (fever, fatigue, muscle aches, shortness of breath, shortness of breath upon exertion, cough, sore throat, stuffy nose, runny nose, loss of taste, loss of smell, headache) by summing the total symptom severities for those symptoms. Higher symptom severities indicates a worse outcome. The minimum and maximum were: 0 to 30, respectively.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
Number analyzed (Participants) | 24 | 23
units on a scale
  Baseline (Day 0) | 16.0000 (6.13614) | 15.5217 (7.21658)
  Day 1 | 14.0417 (6.81736) | 11.0455 (6.26766)
  Day 2 | 12.2500 (6.26411) | 10.0000 (4.98179)
  Day 3 | 11.9583 (6.86186) | 8.6087 (4.09811)
  Day 4 | 10.1667 (6.58501) | 7.7826 (4.79542)
  Day 5 | 9.1667 (5.89522) | 6.0000 (5.03623)
  Day 6 | 7.5417 (5.48499) | 5.3913 (4.39772)
  Day 7 | 7.0417 (5.05173) | 4.6087 (4.56009)
  Day 8 | 6.3333 (5.28054) | 3.9565 (4.17218)
  Day 9 | 6.2500 (5.78040) | 3.6522 (3.92670)
  Day 10 | 5.7917 (5.70262) | 3.0870 (3.08829)
  Day 11 | 5.1667 (6.23919) | 2.4545 (2.72077)
  Day 12 | 4.0000 (6.00000) | 1.9545 (2.57233)
  Day 13 | 4.2083 (5.51661) | 2.0000 (2.39046)
  Day 14 | 4.0417 (6.01071) | 2.1364 (2.41613)
Statistical Analysis 1: Comparison: Modified Qing Fei Pei Du Tang vs Placebo; Test type: Superiority; p = .159, Mixed Models Analysis; F value = 1.987 — day by group interaction

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Modified Qing Fei Pei Du Tang | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/24 | 0/23
Other Adverse Events (participants affected / at risk) | 0/24 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Qing Fei Pei Du Tang (N=24) | Placebo (N=23)
ER visit (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject visited ER due to stomach issues
ER Visit (General disorders) | 1 (1) | 0 (0) — Headache (migraine)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT04939415/Prot_SAP_000.pdf